CLINICAL TRIAL: NCT04729699
Title: Changes and Associations Between Cervical Range of Motion, Pain, Temporomandibular Joint Range of Motion and Quality of Life in Migraineurs Applying Physical Therapy
Brief Title: Changes and Associations Between Cervical Range of Motion, Pain, TMJ Range of Motion and Quality of Life in Migraineurs Applying Physical Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Laura Smilgiene, Laura Smilgiene, physiotherapist, Lithuanian University of Health Science, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2021-01-21; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Migraine; Temporomandibular Joint Disorders; Myofascial Trigger Point Pain
MeSH Terms: conditions — Migraine Disorders; Temporomandibular Joint Disorders; Myofascial Pain Syndromes | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were divided into intervention group and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group (n=10) received 12 physiotherapy sessions and exercises for TMJ 30-45 minutes 2 days per week.
  Interventions: Other: Aerobic exercise and exercise for TMJ
- Control group (Active Comparator): Control group (n=9) was introduced with physiotherapy program in order to perform it independently at home.
  Interventions: Other: Aerobic exercise at home

INTERVENTIONS:
Other: Aerobic exercise and exercise for TMJ — Aerobic exercise
  Arms: Intervention group
Other: Aerobic exercise at home — Aerobic exercise
  Arms: Control group

SUMMARY:
The purpose of this study is to assess the effects of physiotherapy program and review the associations between neck movements, pain, temporomandibular joint (TMJ) movements and quality of life in individuals with migraine.

DETAILED DESCRIPTION:
Migraine is one of the most common type of headaches in the world causing the greatest disability in individuals under 50 years of age. Many different health organizations (American Headache Society etc.) recommend regular physical activity and exercise for the treatment and prevention of migraine. However, the relationship between aerobic exercise and migraine is still not completely clear. Unfortunately, a research database to validate the benefits of exercise for people with migraine is still being developed.

The aim of this study is to assess the effects of physiotherapy program and review the associations between neck movements, pain, temporomandibular movements and quality of life in individuals with migraine.

The study was approved by Committee on Biomedical Research Ethics of Kaunas Region (2020-06-30 No.BEC-SR(M)-266).

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with migraine 2 or more years ago
* Headache, occurring at least 6 times a year
* Individuals from 18 years of age
* Voluntary patient consent to participate in the study

Exclusion Criteria:

* Neurological or psychiatric disorder
* Visiting an orthodontist, taking muscle relaxants
* Head or neck injury, cervical spine hernia, facial or temporomandibular injury

Ages: 37 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
Goniometry for cervical range of motion | Baseline to 6 weeks
  Cervical flexion (45⁰), extension (35⁰) and lateral flexion (45⁰) were measured with mechanical goniometer.
Algometry for pressure pain thresholds (PPT) | Baseline to 6 weeks
  PPT were measured in temporalis, upper trapezius and masticatory muscles with digital algometer in kg/cm²

SECONDARY OUTCOMES:
Anthropometry for TMJ | Baseline and after 6 weeks
  TMJ range of motion was measured with a centimeter before and after physiotherapy
Functional health and well-being - SF-36v2® | Baseline and after 6 weeks
  Quality of life was assessed with the SF-36 questionnaire. Measure is divided into 8 subscales: Physical Functioning, Activity Limitation due to Physical Ailments, General Health, Vitality, Social Functioning, Activity Limitation due to Emotional Problems, General Mental Health and Health Transition. Answers were scored (total score 100) and a higher total score meant a better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Department of Rehabilitation, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided